CLINICAL TRIAL: NCT07152860
Title: Evaluation of the Efficacy of Electroacupuncture in the Treatment of Chronic Atrophic Gastritis: A Randomized Controlled Trial
Brief Title: Evaluation of the Efficacy of Electroacupuncture in the Treatment of Chronic Atrophic Gastritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Liang (Other)
Collaborators: Zhejiang Provincial Department of Science and Technology (Unknown)
Responsible Party: Sponsor-Investigator, Yi Liang, Research Fellow, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250804103318839
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Atrophic Gastritis
Keywords: Chronic atrophic gastritis; electroacupuncture
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture combined with tipronone capsules group (Experimental): Participants will receive acupuncture at seven acupoints: Shangwan(CV13), Zhongwan (CV12) ,Xiawan(CV10), Liangmen (ST21), Tianshu (ST25), Zusanli (ST36), and Xiajuxu (ST39). Disposable needles will be inserted until the "deqi" sensation is achieved. Electroacupuncture is administered at the abdominal points 'CV13-CV12' and 'ST21-ST21', alongside bilateral lower limb points 'ST36-ST39', using an SDZ-IIB handheld electroacupuncture device (Huatuo brand, Suzhou Medical Supplies Factory Co., Ltd.). Receive electroacupuncture treatment at 5Hz.Patients will receive acupuncture treatment three times a week for 1-8 weeks, twice a week for 9-16 weeks, and once a week for 17-24 weeks, for a total of 48 treatments.
  Patients will also be administered SviShu (tipronone capsules) (Wei Cai Pharmaceutical Co., Ltd., National Drug Approval Number H20093656, dosage: 50 mg) orally, one capsule at a time, three times daily, after meals. Treatment will be continued for 24 weeks.
  Interventions: Other: 5 Hz electroacupuncture combined tipronone capsules
- Simple tipronone capsules group(The basic treatment group) (Active Comparator): Patients in the simple tipronone capsules group(basic treatment group) will receive only conventional basic drug therapy. They will be given Svi-Shu (tipronone capsules) (Eisai Pharmaceutical Co., Ltd., national drug approval number H20093656, specification: 50 mg) orally, one capsule at a time, three times a day, after meals. Treatment will be continued for 24 weeks.
  Interventions: Drug: Simple tipronone capsules group(The basic treatment group)

INTERVENTIONS:
Other: 5 Hz electroacupuncture combined tipronone capsules — Intervention Description: The intervention in this study involves the use of electroacupuncture (EA), a combination of traditional acupuncture and electrical stimulation. Acupoints Selection: Electroacupuncture will be performed at specific acupoints associated with the stomach and digestive system. Shangwan(CV13), Zhongwan (CV12) ,Xiawan(CV10), Liangmen (ST21), Tianshu (ST25), Zusanli (ST36), and Xiajuxu (ST39). Disposable needles will be inserted until the "deqi" sensation is achieved. Electroacupuncture is administered at the abdominal points 'CV13-CV12' and 'ST21-ST21', alongside bilateral lower limb points 'ST36-ST39', This selection is based on Traditional Chinese Medicine (TCM) principles for treating chronic atrophic gastritis.
  Frequency: 5 Hz Patients will also be administered SviShu (tipronone capsules) (Wei Cai Pharmaceutical Co., Ltd., National Drug Approval Number H20093656, dosage: 50 mg) orally, one capsule at a time, three times daily, after meals.
  Arms: Electroacupuncture combined with tipronone capsules group
Drug: Simple tipronone capsules group(The basic treatment group) — Patients in the Simple tipronone capsules group(basic treatment group) will receive only conventional basic drug therapy. They will be given Svi-Shu (tipronone capsules) (Eisai Pharmaceutical Co., Ltd., national drug approval number H20093656, specification: 50 mg) orally, one capsule at a time, three times a day, after meals.
  Arms: Simple tipronone capsules group(The basic treatment group)

SUMMARY:
Brief Summary Template for the Study:

This clinical trial aims to evaluate whether electroacupuncture can treat chronic atrophic gastritis (CAG) in adult subjects aged 18 to 75 years (including both males and females), all of whom have been diagnosed with CAG based on endoscopic and histopathological criteria. The primary objectives of this study are to answer the following questions:

* Can 5 Hz electroacupuncture therapy reverse the pathological state of the gastric mucosa in patients with chronic atrophic gastritis?
* Can 5 Hz electroacupuncture therapy improve gastrointestinal symptoms in patients with chronic atrophic gastritis?
* Is there a difference in efficacy between the combination of 5 Hz electroacupuncture therapy and gastric mucosa protectants versus the use of gastric mucosa protectants alone in the treatment of chronic atrophic gastritis?

Researchers will compare the effects of 5 Hz electroacupuncture combined with gastric mucosal protectants versus gastric mucosal protectants alone to determine which method can reverse the pathological state of gastric mucosa and provide more significant symptom relief.

Participants will:

* Receive acupuncture treatment at specific acupoints (such as Shangwan(CV13), Zhongwan (CV12) ,Xiawan(CV10), Liangmen (ST21), Tianshu (ST25), Zusanli (ST36), and Xiajuxu (ST39).) Electroacupuncture is administered at the abdominal points 'CV13-CV12' and 'ST21-ST21', alongside bilateral lower limb points 'ST36-ST39', using an SDZ-IIB handheld electroacupuncture device (Huatuo brand, Suzhou Medical Supplies Factory Co., Ltd.). Receive electroacupuncture treatment at 5Hz.for 30-minute sessions, three times weekly for 1-8 weeks; twice weekly from weeks 9 to 16, once weekly from weeks 17 to 24, for a total of 24 weeks, comprising 48 treatment sessions.
* Be randomly assigned to one of the following groups: 5 Hz electroacupuncture combined with gastric mucosal protective agent group or gastric mucosal protective agent group (control group).
* Have their dyspepsia symptoms, quality of life, and any adverse reactions continuously monitored and assessed throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for chronic atrophic gastritis (CAG) (at the time of enrolment, participants must provide reports from endoscopic and pathological examinations conducted within the past year prior to the study start date, both of which indicate chronic atrophic gastritis)
* Age between 18 and 75 years old, no gender restrictions;
* Has not received acupuncture treatment within the past month;
* Not participated in any other ongoing studies within the past 2 months.
* Understand and agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Autoimmune gastritis (type A chronic atrophic gastritis);
* Participants with a positive C-13 urea breath test at baseline (Helicobacter pylori infection);
* Patients diagnosed with high-grade intraepithelial neoplasia based on upper gastrointestinal endoscopy and gastric mucosal biopsy pathology;
* Patients with confirmed or unresolved malignant tumours, particularly oesophageal cancer and gastric cancer; patients with other upper gastrointestinal lesions such as peptic ulcers or Barrett's oesophagus;
* Patients with severe lesions in major organs (heart, liver, kidney, lung, etc.) or other autoimmune diseases (rheumatic diseases, Crohn's disease, autoimmune pancreatitis, etc.); Persons with cardiac pacemakers;
* Pregnant and lactating women;
* Patients with infectious diseases such as tuberculosis, hepatitis, or HIV/AIDS;
* Individuals with a history of alcohol abuse, drug use, or illicit drug use;
* Individuals who have used other prokinetic agents, mucosal protectants, acid-suppressing medications, or related traditional Chinese medicines within the past two weeks;
* Individuals currently participating in or who have participated in other clinical trials within the past two months; individuals unable to tolerate acupuncture or with contraindications for acupuncture treatment; and individuals deemed unsuitable for participation in this clinical trial by the research team.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Total pathological response rate after 24 weeks of intervention | 24 weeks after the start of treatment.
  Overall reversal rate (%) = (Total number of cases with OLGA or OLGIM reversal after treatment / Total number of cases) × 100% A reversal case is defined as a case where the patient's OLGA or OLGIM stage at week 24 is lower than the baseline stage (a decrease of ≥1 stage in OLGA or OLGIM stage before and after treatment is defined as a reversal, whereas an increase of ≥1 stage is defined as progression). Any stage reversal is counted toward the total number of reversal cases.

SECONDARY OUTCOMES:
Histological scoring of pathological variables | 24 weeks after the start of treatment.
  The histological changes in chronic gastritis include chronic inflammation, active inflammation, atrophy, and intestinal metaplasia, which are classified into four grades: none (0), mild (+), moderate (++), and severe (+++). Each variable is assigned a score based on its grade, with primary variables receiving higher scores: intestinal metaplasia and atrophy at grade 4 are scored as '0, 3, 6, 9 points'; secondary variables receive lower scores: chronic inflammation and activity at grade 4 are scored as '0, 1, 2, 3 points'. The total scores for each variable and the overall pathological score are compared before and after treatment.
Serum pepsinogen I and II (pepsinogen I, pepsinogen II, PG I, PG II), serum pepsinogen ratio (PGR), and gastrin-17 (Gastrin-17) levels. | 24 weeks after the start of treatment.
  Serum pepsinogen levels are an important indicator of dynamic changes in gastric mucosal function. Measurement of PGⅠ, PGⅡ, PGR, and G-17 aids in assessing the extent and severity of gastric mucosal atrophy, and is referred to as 'serological biopsy.' In cases of gastric body atrophy, PGⅠ and PGR levels decrease, while G-17 levels increase; in cases of gastric antrum atrophy, G-17 levels decrease, and the PGⅠ to PGR ratio remains normal; in cases of total gastric atrophy, both levels decrease. Comparisons of serum markers before and after treatment are conducted.
Global Overall Symptom (GOS) Score Change | Baseline, Week 12, Week 24
  The Global Overall Symptom (GOS) score assesses eight symptoms associated with dyspepsia (e.g., epigastric pain, burning, fullness, early satiety, nausea, bloating). Scores range from 1 (no problem) to 7 (very severe problem). Scoring is as follows: 1 = no problem (no symptoms); 2 = minimal problem (can be easily ignored); 3 = mild problem (can be ignored with effort); 4 = moderate problem (cannot be ignored, but does not interfere with daily activities); 5 = moderately severe problem (cannot be ignored, occasionally limits daily activities); 6 = severe problem (cannot be ignored, often limits concentration on daily activities); 7 = very severe problem (cannot be ignored, severely limits daily activities.
Hospital Anxiety and Depression Scale (HADS) Score Change | Baseline, Week 12, Week 24
  The Hospital Anxiety and Depression Scale (HADS) measures levels of anxiety and depression, which are often associated with functional dyspepsia. Changes in HADS scores will be evaluated to determine if electroacupuncture has an impact on emotional well-being. The scores of anxiety and depression subscales are divided into: 0-7 points for no symptoms; 8-10 points for suspected presence; 11-21 points for definite presence; When scoring, 8 points is the starting point, that is, both suspected and symptomatic are positive.
Visual analogue scale (VAS) score for upper abdominal pain | Baseline, Week 12, Week 24
  Assess upper abdominal pain in subjects at weeks 0, 12, and 24. Patients mark the intensity of upper abdominal pain on a straight line from 0 (no pain) to 10 (most severe pain), which is suitable for rapid quantification of subjective pain perception.
Upper abdominal pain diary | Baseline to Week 24
  Patients should record the frequency, duration, triggering factors (e.g., eating, stress), and accompanying symptoms (e.g., nausea, acid reflux) of each episode of upper abdominal pain during the entire treatment period. They should also record the types and doses of medications used to relieve upper abdominal pain (e.g., antacids, acid suppressants, antispasmodics, traditional Chinese medicines, etc.).
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 12, Week 24
  Assess the PSQI scores of the subjects at weeks 0, 12, and 24. This scale is the most commonly used scale for evaluating sleep quality in recent years. A PSQI score > 7 is considered to indicate poor sleep quality, while a PSQI score ≤ 7 is considered to indicate good sleep quality.
Treatment Expectation Score | Prior to the first treatment (Baseline)
  Before treatment, patients are asked to assess their expectations of the efficacy of electroacupuncture. Patients are asked to evaluate the efficacy of electroacupuncture (electroacupuncture treatment will significantly improve my pathological condition) using a five-point scale: 'strongly agree,' 'somewhat agree,' 'neutral,' 'somewhat disagree,' and 'strongly disagree.' This is done to collect patients' expectations of electroacupuncture treatment.
Compliance evaluation | Baseline, Week 12, Week 24
  Assess whether subjects at weeks 12 and 24 completed treatment and questionnaire collection at that point in time. If there are any withdrawals, exclusions, or dropouts during the study, promptly record the time of study termination and the specific reasons for termination.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Hangzhou TCM Hospital of Zhejiang Chinese Medical University (Hangzhou Hospital of Traditional Chinese Medicine), Hangzhou, Zhejiang
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The Third Affiliated Hospital of Zhejiang Chinese Medicinal University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF